## Cover Page

Study Title: Homeless Youth Study - Stepping Stone 2.0

Document Type: Study Protocol with Statistical Analysis Plan (SAP)

Document Date: 11/5/2018

## **Study Protocol**

The study will take 3-6 months and will consist of the following:

- Participants will complete a 1.5 hour enrollment session including the informed consent process, self-report questionnaires, phone set-up, and a phone usage and safety briefing.
- Over the course of 3 months, participants will have access to automated self-help interventions designed as a kit of smartphone tools, which are based on principles of cognitive-behavioral therapy. Participants will also have access to three services that will connect them with a real person if they need emotional support.
- Participants will have the opportunity to complete two optional 30-minute interviews at 2 weeks and 4 weeks into the study period.
- Participants will also be asked to complete a daily survey and rate a daily tip via a mobile app.
- At the 3-month point of the intervention, participants will be asked to complete another series of self-report questionnaires. If these questionnaires are completed with valid responses, participants will receive another 3 months of paid phone service and study participation will be extended to 6 months.
- At the end of the 6-month period, participants will be asked to complete an endpoint assessment consisting of self-report questionnaires. A \$25 incentive will be offered for completing this assessment.

## Statistical Analysis Plan

- We will examine usage of the mobile applications, ratings of acceptability, and ratings of perceived benefit.
- We will conduct paired t-tests to assess pre-post change in posttraumatic stress disorder, depression, anxiety, substance use, risky behaviors, satisfaction with life, and psychosocial flourishing.